CLINICAL TRIAL: NCT05306990
Title: Efficacy and Safety of Atorvastatin 40mg Versus Rosuvastatin 20mg in Type II Diabetic Patients With Previous Acute Coronary Syndrome : Randomized Clinical Trial
Brief Title: Statins in Patients With Type 2 Diabetes Mellitus and Previous History of Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Yassmin Genina, Teaching assistant at pharmacy practice department Faculty of pharmacy Helwan University, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pharmacy practice department
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Hydroxymethylglutaryl-CoA Reductase Inhibitors; Diabetes Mellitus
Keywords: High intensity statin therapy; Acute coronary syndrome; Atorvastatin; Rosuvastatin; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Acute Coronary Syndrome | interventions — Atorvastatin; Tablets; ORANGE protein, Arabidopsis; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Active Comparator): Atorvastatin tablets Dosage and frequency: 40mg orally once daily
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet
- Rosuvastatin (Active Comparator): Rosuvastatin tablets Dosage and frequency: 20mg orally once daily
  Interventions: Drug: Rosuvastatin 20 Mg Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — patients followed up for 3 months
  Other Names: Ator
  Arms: Atorvastatin
Drug: Rosuvastatin 20 Mg Oral Tablet — patients followed up for 3 months
  Other Names: crestor
  Arms: Rosuvastatin

SUMMARY:
The purpose of this study was to compare the efficacy and safety of high dose atorvastatin (40 mg) versus high dose rosuvastatin (20 mg) in Egyptian type II diabetic patients with previous acute coronary syndrome history. This open-labeled prospective, randomized clinical trial compared once daily atorvastatin 40mg (Ator®) versus once daily rosuvastatin 20mg (Crestor®). The primary outcome was the 50% reduction in low-density lipoprotein cholesterol levels at 12 weeks. The secondary outcome was the achievement of low-density lipoprotein cholesterol level < 55 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis with type 2 diabetes.
* Previous history of acute coronary syndrome.
* Abnormal baseline lipid profile.

Exclusion Criteria:

* Patients taking concurrent lipid lowering agents such as bile acid sequestrants (cholestyramine, colesevelam), niacin, ezetimibe, fenofibrate and/or omega3.
* Patients taking concurrent interacting medications such as ciclosporin, gemfibrozil, clarithromycin and/or itraconazole.
* Patients with active liver disease, bile duct problems, or ALT > 3 × upper limit of normal (ULN).
* Patients with serum creatinine > 2 mg/dl.
* Patients have incidence or history of hypersensitivity reaction to any of the statin used.
* Women who were pregnant, breast-feeding or of child-bearing potential and not using a reliable form of contraception at the time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Mean Change from baseline in Low Density Lipoprotein Cholesterol (LDL-C) | Post intervention at week 12
  A measure of participants with response

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No